CLINICAL TRIAL: NCT04088838
Title: Natural Course of Pain Following Surgery Through an Abdominal Incision: The Role of Adhesions and Other Factors in Chronification of Abdominal Pain
Brief Title: Natural Course of Pain Following Surgery Through an Abdominal Incision
Acronym: Pain Trac
Status: Active, not recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-5241; NL68853.091.19 (Registry Identifier: CCMO register (Dutch ethical approval register))
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Adhesions Abdominal; Adhesions Pelvic; Surgery Induced Tissue Adhesions; Chronic Pain
MeSH Terms: conditions — Tissue Adhesions; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing abdominal surgery: All adult patients undergoing elective abdominal surgery are eligible. Abdominal surgery includes each operation in which the peritoneal cavity is openen, i.e. laparotomy or laparoscopy.
  Interventions: Other: Pain tracking app

INTERVENTIONS:
Other: Pain tracking app — In this study no clinical interventions are made. Patients scheduled for surgery will be treated according to the standard of care. All patients enrolled will have an application installed to track their pain symptoms through short daily and weekly questionnaires.

SUMMARY:
Chronic abdominal pain is highly prevalent in patients undergoing abdominal surgery. Adhesions are reported to be one of the most common causes of chronic pain after surgery. There is little epidemiological data on the natural course and risk factors of pain. In this study the investigators will assess risk factors for chronic pain and natural course by tracking pain scores through an app in a cohort of 1,500 patients undergoing abdominal surgery. In part two of the study patients with persistent abdominal pain at 12 months, that meet IASP criteria for chronic pain will have clinical investigations to determine the cause of their pain. This investigation includes cineMRI for diagnosis and mapping of adhesions.

DETAILED DESCRIPTION:
Rationale: Chronic abdominal and pelvic pain are highly prevalent in among patients who had abdominal surgery in history. An estimate of 11-20% of all patients undergoing different kinds of abdominal surgery will develop chronic abdominal pain. Adhesions (a form of internal scar tissue) are the most common pathology found in patients undergoing diagnostic laparoscopy for pain. Other factors that might be associated with chronic post-operative pain are anxiety, depression, and female sex. Little is known about the natural course of pain after abdominal surgery, risk factors for developing chronic pain, and the mechanisms causing pain in patients with adhesions. In this longitudinal study the investigators will prospectively study the natural course of pain through repeated measurements, and predictive factors for chronification of pain after different types of abdominal surgery.

Objective: In Phase 1 the investigators will study the natural course of pain following abdominal surgery. Primary objective for phase 1 is to assess risk factors for chronic pain at 12 months after surgery; where chronic pain is defined as daily continues or intermittent pain with maximal pain scores of 4 or higher during more than 3 months in accordance to IASP criteria. As a pivotal secondary outcome we will describe and model the duration (days) of moderate (worst pain score 4 to 6) to severe pain (worst pain score 7 or higher), and assess factors that impact the chance in painscore using mixed models. In phase two the investigators will assess the impact of adhesions on chronic pain. Primary objective for phase two is to compare incidence and extent of adhesions on cineMRI between patients who developed chronic pain and patients who did not develop chronic pain at 12 months after surgery.

Study design: This is prospective cohort study, including 1,500 patients scheduled for elective abdominal surgery. In phase one, patients are asked to fill a comprehensive questionnaire, including quality of life assessment and a comprehensive assessment of potential predictive factors for chronic pain prior to surgery. Post-operatively pain symptoms will be monitored using short daily and weekly questionnaires taken by m-health and e-health techniques to study natural course of pain. A comprehensive assessment of pain, quality of life, and medical consumption will be taken at 3,6, and 12 months post-operatively.

In phase two of the study patients who developed chronic pain will be invited for mapping of adhesions using cineMRI. Results of mapping of adhesions using cineMRI in patients with chronic abdominal pain will be compared to mapping of adhesions in 100 patients matched for type of surgery and risk factors who did not develop chronic pain.

Study population: 1,500 patients undergoing elective abdominal surgery from different surgical subspecialties (e.g. colorectal, upper-GI, and gynaecological surgery), aged 18 years or older.

Main study parameters/endpoints: Main study outcome for phase one are risk factors for development of chronic pain at 12 months post-operative. Pivotal secondary outcomes include description of the median duration (days) of moderate to severe abdominal pain following abdominal surgery, and modelling of factors that impact change in abdominal pain after surgery. Other secondary outcomes include health-related quality of life, healthcare utilization, and return to daily activity or work.

Main outcomes for phase two is the percentage of patients with adhesions on cineMRI as compared between patients with and without chronic pain. Secondary outcomes relate to the appearance of adhesions on cineMRI, and included extent and the loss of shear.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In phase one of this cohort study patients will be asked to fill repeated questionnaires on pain and potential risk factors for chronic pain. The intake questionnaire prior to surgery will take approximately 60 minutes to fill. Post-operatively we will send short questionnaires that take 2-5 minutes to fill. These questionnaires will be send daily during the first 60 days after surgery and weekly afterwards. A more comprehensive questionnaire on abdominal pain and complaints that takes 45 minutes to complete will be send at 3,6, and 12 months post-operative. There are no risks related to participation in this study, nor are there direct benefits.

Patients participating in part two of this cohort will undergo cineMRI to evaluate if pain symptoms might relate to adhesions form previous surgery. The MRI will take approximately 20 minutes to perform. MRI is a non-invasive imaging technique without health risks. However, there is a risk of incidental findings that do not relate to the subject of this study (adhesion formation). Patients who do not want to be informed about incidental findings will be excluded from phase two. In a subset female patients who had pelvic surgery and resection of the uterus an additional transvaginal ultrasound will be made. Like MRI, this is a non-invasive diagnostic test without health risks. There is some additional inconvenience by the use of a transvaginal ultrasound prove. The test will take approximately 15 min.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Adult patients, aged above 18 years
* Planned for elective abdominal surgery, e.g. laparotomy or laparoscopy

For phase two of this study we will recruit patients from the group that participated in phase 1. Additional inclusion criteria for phase two:

* Patients who developed chronic post-operative abdominal pain according to IASP criteria:
* Daily pain in the past three months
* Pain is continues or intermittent
* Pain scores for the worst pain are 4 or higher
* Or patients without chronic pain (n=100) who are propensity matched for type of surgery and risk factors for developing chronic pain.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Mental incompetence
* Planned for laparoscopic cholecystectomy
* Planned for Caesarean section

Additional exclusion criteria for phase two are:

* Contra-indications for MRI (without contrast) including:
* Severe claustrophobia
* Metal splinters in eyes
* Cerebral vascular clips
* Electronic medical implants
* Patients who do not want to be informed about potential incidental findings of MRI-scan

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with undergoing different types of abdominal surgery (laparotomy and laparoscopy). Included are all patients undergoing elective surgery. Patients undergoing laparoscopic cholecystectomy and caesarean section are excluded because both are very frequent procedures with a low risk of chronic post-operative pain and low risk of adhesions. These procedure could therefore significantly impact the power of the study. Although patients after laparoscopic cholecystectomy frequently report pain, these pain symptoms are often attributable to persistence of pre-existing pain. There are known difficulties in differential diagnosis of symptomatic cholelithiasis and dyspepsia, that might interfere with indication for cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Risk factors for development of chronic pain | 12 months
  Prediction model for development of chronic post-operative abdominal pain, assessed using a dynamic prediction model. Potential factors are taken from baseline measurements, and the repeated measurements of the course of pain.
Incidence of adhesions on cineMRI in patients with chronic abdominal pain. | 2 months
  Primary outcome of the second phase of study in which patients with chronic pain will undergo clinical investigations determining the cause of their pain,

SECONDARY OUTCOMES:
incidence of chronic pain | 12 months
  Descriptives of incidence of chronic pain at 12 months post-operative
Duration of moderate to severe pain | 60 days post surgery
  duration of moderate (worst pain score 4 to 6) to severe (worst pain score 7 or higher) following abdominal surgery
Health-related quality of life | 12 months
  EuroQol Q5-5D-5L
Return to daily activity/ work | 12 months
  measured by iPCQ
Healthcare utilization | 12 months
  measured by iMCQ
characteristics of adhesions on cineMRI | 2 months
  Descriptives of appearencesuch as extent, loss of shear, organ involvement

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Maasziekenhuis Pantein, Boxmeer, Gelderland
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Maastricht Universitair Medisch Centrum+, Maastricht, Limburg
  - Rijnstate Hospital, Arnhem
  - Slingeland Hospital, Doetinchem
  - Gelderse Vallei Hospital, Ede
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study a copy of the data will be stored in DANS easy archive. Anonymized data will be made available for other researcher 2 years after completion of the study and upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years after completion of the study. No time limit is associated with storage of data in the aforementoined archive.
Access Criteria: Data will be made available upon reasonable request. Request will be evaluated by the steering group of the study. Request will be granted when meeting the following criteria:
  * Analysis plan meeting requirements as set by Dutch law and regulations for medical research and privacy.
  * Data is made available for the research question as proposed in the analysis plan.
  * The research question has not posed previously by the steering groups or in another request.
  * A timeframe during which analysis will be performed will be areed upon. If analysis is not completed within this time frame, the steering group might make the data available again to other researcher for this research question.
  * depending on the research question the steering group might propose to be involved as co-authors
  * In case of data request from researchers of a commercial party additional criteria might apply

REFERENCES:
- [Background] van den Beukel BAW, Stommel MWJ, van Leuven S, Strik C, IJsseldijk MA, Joosten F, van Goor H, Ten Broek RPG. A Shared Decision Approach to Chronic Abdominal Pain Based on Cine-MRI: A Prospective Cohort Study. Am J Gastroenterol. 2018 Aug;113(8):1229-1237. doi: 10.1038/s41395-018-0158-9. Epub 2018 Jun 27. PMID 29946174
- [Background] Strik C, van den Beukel B, van Rijckevorsel D, Stommel MWJ, Ten Broek RPG, van Goor H. Risk of Pain and Gastrointestinal Complaints at 6Months After Elective Abdominal Surgery. J Pain. 2019 Jan;20(1):38-46. doi: 10.1016/j.jpain.2018.07.010. Epub 2018 Aug 11. PMID 30107242
- [Background] Randall D, Joosten F, Ten Broek RP, Gillott R, Bardhan KD, Strik C, Prins W, van Goor H, Fenner JW. A novel diagnostic aid for intra-abdominal adhesion detection in cine-MRI: pilot study and initial diagnostic impressions. Br J Radiol. 2017 Aug;90(1077):20170158. doi: 10.1259/bjr.20170158. Epub 2017 Jul 14. PMID 28707532
- [Background] van den Beukel BA, de Ree R, van Leuven S, Bakkum EA, Strik C, van Goor H, Ten Broek RPG. Surgical treatment of adhesion-related chronic abdominal and pelvic pain after gynaecological and general surgery: a systematic review and meta-analysis. Hum Reprod Update. 2017 May 1;23(3):276-288. doi: 10.1093/humupd/dmx004. PMID 28333221